CLINICAL TRIAL: NCT03783728
Title: Efficacy of Risk-Targeted Video Based Directly on Observed Therapy for Latent TB
Brief Title: Video Based Directly Observed Therapy for Latent TB
Status: Withdrawn | Type: Observational
Why Stopped: Investigator is leaving the University
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Soumya Chatterjee, MD, Assistant Professor of Internal Medicine, St. Louis University
Other Study IDs: 29312
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Latent Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis | interventions — rifapentine; Isoniazid; Pyridoxine; Vitamin B 6

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 20 mL of Peripheral Blood Mononuclear Cells (PBMCs) will be collected for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

GROUPS / COHORTS (1):
- Untreated Latent Tuberculosis Infection: Isoniazid 900 mg orally + Rifapentine 600 mg orally + Pyridoxine 50 mg orally once a week for 12 weeks
  Interventions: Drug: Rifapentine 600 mg orally; Drug: Isoniazid 900 mg orally; Drug: Pyridoxine 50 mg orally

INTERVENTIONS:
Drug: Rifapentine 600 mg orally — Once a week for 12 weeks using Video Directly Observed Therapy
  Other Names: Priftin
Drug: Isoniazid 900 mg orally — Once a week for 12 weeks using Video Directly Observed Therapy
  Other Names: INH
Drug: Pyridoxine 50 mg orally — Once a week for 12 weeks using Video Directly Observed Therapy
  Other Names: Vitamin B6

SUMMARY:
Center for Disease Control (CDC) data reveal that after years of sustained decrease, the incidence of active tuberculosis (TB) disease in the US has plateaued. Most of the cases occur when Mycobacterium tuberculosis (Mtb) reactivates replication in people who have latent tuberculosis infection (LTBI). Only 5 to 10% of subjects with LTBI develop active TB Infection over their lifetime. Current US guidelines recommend treating everyone with LTBI to stop progression to active TB. As treatment is long, only about 45-55% of patients finish treatment overall, regardless of whether the patients are at high (>10%) or low lifetime risk of reactivation. The investigator's study aims to test the efficacy of a combined approach of first determining subjects at high risk of reactivation and then treating them with a CDC approved once a week treatment regimen, directly observed by a nurse over video (video-based Directly Observed Therapy, vDOT). Ensuring treatment of the high-risk group will eventually decrease the community active TB burden.

DETAILED DESCRIPTION:
Tuberculosis (TB) in the US: Tuberculosis (TB), caused by the bacterium Mycobacterium tuberculosis (Mtb), is a leading cause of mortality, killing more than a million people worldwide^1. In the United States an important recent trend has been the plateauing of the active TB disease incidence at 3.0 cases per 100,000 persons^2. Current US TB control guidelines recommend treating all subjects with LTBI to prevent progression to active TB. However, treatment is given with the antibiotic Isoniazid (INH) for 6-9 months, Rifampin and Rifabutin for 4 months or INH with Rifapentine for 3 months and as subjects with LTBI are asymptomatic, treatment default rates are understandably high (>10% on average)^3-5. It is well known that a subset of patients with LTBI have higher risk of progression to active TB. Because of the high treatment default rate, a number of these "high risk" subjects receive incomplete or no preventive therapy and contribute to the incidence of active TB cases in the US. Currently, there are no strategies being implemented to identify those at highest risk and consequently treatment approaches follow the "one size fits all" paradigm. In the investigators preliminary study done at the Saint Louis University (SLU) Infectious Diseases Clinic, the investigators used an online risk calculator (TSTin3D.com)^6 to retrospectively determine the cumulative lifetime risk of progression to active TB for adults receiving treatment for latent TB. The investigators found that current practice leads to equal rates of treatment completion i.e. 57% in the high risk for active TB disease (TBhi) group (>10% cumulative risk of progression based on medical risk factors) compared to 59% for those at lowest risk (TBlow, <10% cumulative risk of progression). It is not standard of care to use a scoring system like the TSTin3d.com to assess the risk. There are certain risk factors like having HIV or being on immunosuppression that physicians ask about but most physicians do not do a quantitative risk assessment. Treatment choices are usually based on convenience and concern for side effects but the most common regimen is daily INH for 6-9 months.

This data implies that the current "treat everyone and hope that therapy is completed" approach leads to a significant number of people in the TBhi group remaining untreated and at high risk of progression to active TB. A recent advance has been a CDC approved regimen using Isoniazid (INH) and Rifapentine given weekly as directly observed therapy (DOT) for 12 weeks (known as the 3HP regimen). This regimen has shown lower toxicity, better adherence and equivalent efficacy^7-12. INH + Rifapentine (3HP) is not currently used widely as DOT is resource intensive. The investigators hypothesize that if providers use the calculator (TSTin3d.com) to firstly determine risk and then select the once weekly DOT for the TBhi group (12 doses total); the investigators can ensure that the TBhi group completes treatment. Complete treatment of the TBhi group will have the highest impact in decreasing the community burden of TB disease. The investigators propose the first US study to prospectively test the efficacy of an approach which 1) defines the TBhi group using TSTin3d.com and 2) ensures treatment completion in the TBhi group with weekly with video-based DOT (vDOT) with 3HP. Most patients nowadays have access to a smartphone with video capabilities. A HIPAA approved video application (Zoom) is already available through the Missouri Telehealth Network and can be used by the patient to interface with the TB clinic nurse over a smartphone. The investigators approach removes the need for the patients in the TBhi group to be physically present in the TB clinic. All patients identified in the TBhi group can thus be safely provided vDOT. The investigators pilot study has important implications for improving care and patient treatment outcomes as it will identify the "high risk" subjects with latent TB using tstin3d.com (Table 1), [a validated online calculator that combines TST or interferon Gamma Release Assay (IGRA) screening results with clinical information obtained from the patient, to generate an individual's cumulative risk of developing active TB disease, up to age 80^11]. The investigators will then ensure that patients complete therapy under direct observation by a nurse using video based Directly Observed Therapy (vDOT). vDOT also eliminates the need for the patient to physically visit the clinic. All patients need is access to a smartphone with video capabilities. HIPAA approved video based applications are already available for vDOT and has already been implemented successfully.^13

All of the drug options listed are standard of care currently in the US. It is currently not standard of care to use a scoring system like tstin3d.com to assess risk. There are certain risk factors like having HIV or being on immunosuppression that physicians routinely ask about but most physicians do not do a quantitative risk assessment. Treatment choices are usually based on convenience and concern for side effects but the most common regimen is daily INH for 6 months or 9 months.

ELIGIBILITY:
Inclusion Criteria:

- Age 18 years + 1 day (defined as date of birth plus one day). This age cutoff has been selected as tstin3d.com has only been validated for this age group.

Subjects must have all of the following:

* Untreated Latent Tuberculosis Infection (LTBI), defined as positive Tuberculin skin test/QuantiFERON TB Gold test or T-spot assay done within 1 month prior to enrollment.
* Absence of active TB disease as determined by history, physical examination, chest X-ray, (sputum smear and/or culture done as needed by the assessing physician for Mtb).
* Greater than 10% cumulative risk of developing active TB disease (determined by TSTin3D.com).

Exclusion Criteria:

* A subject will be excluded if any of the following criteria are met:
* Presence of active TB disease
* BMI <16
* Cardiovascular instability (Blood pressure: Systolic >180 or <90 mm/Hg or Diastolic >100 or < 50mm/Hg; pulse <40 or >110)
* Chest X-Ray report within last 3 months not available
* HIV positive and currently on treatment with a regimen that has severe drug interactions with 3HP.
* Presumed infected with INH or Rifapentine (RIF)-resistant M. tuberculosis
* Women who are pregnant, nursing or expect to become pregnant for the duration of the study.
* Temperature ≥38.5°C or other clinical evidence of an acute infection at screening
* History of treatment for >14 consecutive days with a rifamycin or >30 consecutive days with isoniazid during the previous 2 years
* Documented history of completing adequate treatment for active tuberculosis or latent M. tuberculosis infection in a HIV-seronegative person
* History of sensitivity/intolerance to isoniazid or rifamycins
* Serum aspartate aminotransferase (AST) >5 times the upper limit of normal (ULN) if AST was determined
* Hemodynamic instability or medical/psychological condition precluding participation in the study as judged by the investigator
* No access to a smartphone for personal use
* Refuse blood draws
* Refuse to participate in the study
* If female of childbearing potential and on a hormonal contraception method, refuse to use an additional barrier method with the hormonal method for the duration of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with latent tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-30 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients completing treatment | 4 months
  Achieving > 90% treatment completion in patients with LTBI at > 10% cumulative individual risk of developing active TB using vDOT.

CONTACTS AND LOCATIONS:
Overall Officials: Soumya Chatterjee, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

REFERENCES:
- [Result] Salinas JL, Mindra G, Haddad MB, Pratt R, Price SF, Langer AJ. Leveling of Tuberculosis Incidence - United States, 2013-2015. MMWR Morb Mortal Wkly Rep. 2016 Mar 25;65(11):273-8. doi: 10.15585/mmwr.mm6511a2. PMID 27010173
- [Result] Li J, Munsiff SS, Tarantino T, Dorsinville M. Adherence to treatment of latent tuberculosis infection in a clinical population in New York City. Int J Infect Dis. 2010 Apr;14(4):e292-7. doi: 10.1016/j.ijid.2009.05.007. Epub 2009 Aug 4. PMID 19656705
- [Result] Stuurman AL, Vonk Noordegraaf-Schouten M, van Kessel F, Oordt-Speets AM, Sandgren A, van der Werf MJ. Interventions for improving adherence to treatment for latent tuberculosis infection: a systematic review. BMC Infect Dis. 2016 Jun 8;16:257. doi: 10.1186/s12879-016-1549-4. PMID 27268103
- [Result] Sterling TR, Scott NA, Miro JM, Calvet G, La Rosa A, Infante R, Chen MP, Benator DA, Gordin F, Benson CA, Chaisson RE, Villarino ME; Tuberculosis Trials Consortium, the AIDS Clinical Trials Group for the PREVENT TB Trial (TBTC Study 26ACTG 5259) The investigators of the TB Trials Consortium and the AIDS Clinical Trials Group for the PREVENT TB Trial are listed in the Supplement, item 17. Three months of weekly rifapentine and isoniazid for treatment of Mycobacterium tuberculosis infection in HIV-coinfected persons. AIDS. 2016 Jun 19;30(10):1607-15. doi: 10.1097/QAD.0000000000001098. PMID 27243774
- [Result] Sterling TR, Moro RN, Borisov AS, Phillips E, Shepherd G, Adkinson NF, Weis S, Ho C, Villarino ME; Tuberculosis Trials Consortium. Flu-like and Other Systemic Drug Reactions Among Persons Receiving Weekly Rifapentine Plus Isoniazid or Daily Isoniazid for Treatment of Latent Tuberculosis Infection in the PREVENT Tuberculosis Study. Clin Infect Dis. 2015 Aug 15;61(4):527-35. doi: 10.1093/cid/civ323. Epub 2015 Apr 22. PMID 25904367
- [Result] Bliven-Sizemore EE, Sterling TR, Shang N, Benator D, Schwartzman K, Reves R, Drobeniuc J, Bock N, Villarino ME; TB Trials Consortium. Three months of weekly rifapentine plus isoniazid is less hepatotoxic than nine months of daily isoniazid for LTBI. Int J Tuberc Lung Dis. 2015 Sep;19(9):1039-44, i-v. doi: 10.5588/ijtld.14.0829. PMID 26260821
- [Result] Sterling TR, Villarino ME, Borisov AS, Shang N, Gordin F, Bliven-Sizemore E, Hackman J, Hamilton CD, Menzies D, Kerrigan A, Weis SE, Weiner M, Wing D, Conde MB, Bozeman L, Horsburgh CR Jr, Chaisson RE; TB Trials Consortium PREVENT TB Study Team. Three months of rifapentine and isoniazid for latent tuberculosis infection. N Engl J Med. 2011 Dec 8;365(23):2155-66. doi: 10.1056/NEJMoa1104875. PMID 22150035
- [Result] Holzschuh EL, Province S, Johnson K, Walls C, Shemwell C, Martin G, Showalter A, Dunlay J, Conyers A, Griffin P, Tausz N. Use of Video Directly Observed Therapy for Treatment of Latent Tuberculosis Infection - Johnson County, Kansas, 2015. MMWR Morb Mortal Wkly Rep. 2017 Apr 14;66(14):387-389. doi: 10.15585/mmwr.mm6614a3. PMID 28406884
- [Result] Menzies D, Gardiner G, Farhat M, Greenaway C, Pai M. Thinking in three dimensions: a web-based algorithm to aid the interpretation of tuberculin skin test results. Int J Tuberc Lung Dis. 2008 May;12(5):498-505. PMID 18419884
- See also: World Health Organization (WHO) TB Report — http://who.int/tb/publications/global_report/en/.